CLINICAL TRIAL: NCT05276960
Title: A Randomized, Double-blind Study of the Efficacy of Intensive Cholecalciferol Monitoring and Supplementation on Serum Vitamin D Levels in Pediatric Patients With Cystic Fibrosis
Brief Title: Efficacy of Intensive Cholecalciferol Monitoring and Supplementation on Serum vitD Levels in Pediatric Patients With CF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Magali Reyes Apodaca, Principal Investigator, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIM-2021-087
Record Dates: First submitted 2022-02-21; First posted 2022-03-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Vitamin D Deficiency; Cystic Fibrosis; Bone Density, Low; Inflammation Chronic; Cystic Fibrosis in Children; Cystic Fibrosis Pulmonary Exacerbation
Keywords: vitamin D; cystic fibrosis; pulmonary exacerbation; Vitamin D Deficiency or insufficiency
MeSH Terms: conditions — Vitamin D Deficiency; Cystic Fibrosis; Bone Diseases, Metabolic | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Pediatric CF patients will be recruited from the CF Integrated Care Clinic of the Federico Gomez Children's Hospital of Mexico. Once at the clinic they will be invited to participate in the study. Parents or guardians of patients under 8 years of age will be asked to sign the informed consent form before starting the studies, procedures and intervention. For those patients older than 8 years, in addition to parental consent, they will be given information and asked to sign the informed consent form before starting the studies, procedures, and intervention.
  The restrictive randomization will be performed by blocks of 8,obtained through the web page https://www.randomizer.org/, and will be carried out by one of the investigators, who will also be responsible for its safekeeping. The concealment will be carried out by the same investigator in charge of the randomization, for which the treatment groups will be placed in metallic gray, non-transparent, previously labeled envelopes
Who Masked: Participant, Care Provider, Investigator
Masking Description: For the blinding of the maneuver, supplementation will be done with cholecalciferol (vitD3) in dispersible tablets of the same size and color, with doses of 2000 IU (0.05 mg) for the control group and 4000 IU (0.1 mg) for the intervention group. The capsules should be dissolved in 30 ml of water. The dispensing of the medication according to the intervention group and vitamin D levels will be performed by the investigator assigned to blinding of the principal investigator, the containers of the tablets will be of the same color and size and only the investigators responsible for the dispensing will know the corresponding dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regular supplementation (Active Comparator): Baseline dose of 2000 IU of vitamin D3, based on Cystic Fibrosis Foundation (CFF) treatment guidelines. According to serum vitamin D levels, 2000 IU increments will be performed whenever 25-OH-VitD (25-hydroxy vitamin D) values < 30 ng/ml are found.
  Interventions: Drug: Cholecalciferol Pill
- Enhanced Supplementation (Experimental): Basal dose of 4000 IU of vitamin D3. According to serum vitamin D levels, increments of 4000 IU will be made each time 25-OH-VitD values < 30 ng/ml are found.
  Interventions: Drug: Cholecalciferol Pill

INTERVENTIONS:
Drug: Cholecalciferol Pill — Dose increments according to serum levels determined every 2 months

SUMMARY:
Cystic fibrosis (CF) is an autosomal recessive disease caused by alterations in the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) gene, characterized by multisystemic alterations, mainly in the lung, intestine, sweat, and bile ducts. In addition to pulmonary involvement, the presence of exocrine pancreatic insufficiency also increases the risk of survival, as it is associated with malnutrition and deficiency of fat-soluble vitamins, such as vitamin D.

Vitamin D, in addition to its role in bone health, in the case of CF patients with chronic inflammation, it has been suggested that many of the cytokines that regulate the inflammatory response contain elements that respond to vitamin D, so vitamin D could play an essential role in the regulation of the inflammatory response in CF, which could favor lung function.

However, more than 50% of CF patients present vitamin D insufficiency or deficiency, despite the different schemes suggested for supplementation in different age groups, which suggests that new strategies are needed to normalize vitamin D levels, which will allow us to see its clinical effect on the inflammatory response, by decreasing the number of exacerbations and thus perpetuating or improving lung function, as well as on bone mineral health.

DETAILED DESCRIPTION:
Randomized double-blind clinical trial in patients aged 5 to 18 years attending the CF Comprehensive Care clinic in Mexico City. The intervention group will receive an intensification of vitamin D supplementation, with increments of 4000 IU depending on serum levels, the control group will receive supplementation according to the treatment guidelines of the Cystic Fibrosis Foundation, and the dose will be doubled depending on serum levels. In both groups vitamin D levels will be measured at 3, 6, 9, and 12 months, spirometry and sputum culture will also be performed to evaluate the pulmonary function, densitometry to evaluate the bone mineral density and body composition, together with anthropometric evaluation and quantitative bone ultrasound at each visit, in the biochemical evaluation, calcium/creatinine ratio and alkaline phosphatase will be taken at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis

Exclusion Criteria:

* Another chronic disease (HIV, cancer, renal failure)
* 25-OH-VitD levels < 10 ng/ml or > 30 ng/ml

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in VitD Levels | Baseline, every 2 months through study completition, an avarage of 1 year.
  Serum vitamin D levels up to 30 ng/ml

SECONDARY OUTCOMES:
Changes in the number of Pulmonary exacerbations | 12 months
  Number of exacerbations present during 1 year prior and 1 year after the baseline
Changes in the Bone mineral density | 12 months
  changes in bone mineral content at baseline and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Magali R Reyes Apodaca, MSc, Principal Investigator — Hospital Infantil de Mexico Federico Gomez; Mara Medeiros, MD, Msc, PhD, Study Director — Hospital Infantil de Mexico Federico Gomez
Locations (1):
- Hospital Infantil de México Federico Gómez, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No